CLINICAL TRIAL: NCT01578993
Title: A Phase IV, Prospective Clinical Evaluation of Complications Related to the Use of Peripherally Inserted Central Catheters (PICC) - An Observational Baseline Multicenter Study.
Brief Title: Observational Study of Complications Related to Use of Peripherally Inserted Central Catheters
Acronym: PRISM-1
Status: Completed | Type: Observational
Sponsor: Teleflex (Industry)
Responsible Party: Sponsor
Other Study IDs: S-PICC 2012-01
Record Dates: First submitted 2012-04-12; First posted 2012-04-17 (Estimated); Results first posted 2014-06-24 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2014-05

CONDITIONS: Adult Patients With Peripherally Inserted Central Catheters

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the rate and timing of interventions and complications related to the use of peripherally inserted central venous catheters in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female Age > 18 years requiring central venous access
* Ability to comply with study requirements
* Written Informed Consent

Exclusion Criteria:

* Previous enrollment in study
* Current or recent upper extremity thrombosis, occlusion or stenosis
* Previous axillary lymph node dissection
* Skin inflammatory condition or rashes within 15 cm from insertion site
* Pre-existing history of hypercoagulability unrelated to malignant disease
* Participating in trial involving antithrombotic, anticoagulant or anti- infective drug therapies
* Positive blood culture within 48 hours from planned PICC placement
* Known, renal insufficiency with chronic creatinine levels > 1.7 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients necessitating insertion of a PICC for fluid, nutritional, chemotherapy or antibiotic treatment for a minimum of 14 days.
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ronald Reagan UCLA Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Study: Patients requiring a standard 5 Fr Dual Lumen Peripherally Inserted Central Catheter (PICC) for an anticipated minimum 14 Days of antibiotic, chemotherpay or nutritional support were eligible for enrollment into this observational study.
Period: Overall Study
Arm/Group | Single Arm Study
Started | 101
Completed | 101
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Study
Number analyzed (Participants) | 101
Age, Continuous [Median (Full Range); unit: Years] | 55 [18 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 7
  White | 88
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 101

OUTCOME MEASURES:

1. Primary Outcome: Rate of PICC Line Occlusions
Description: The incidence, severity and management of PICC line occlusions were recorded for each of the enrolled subjects.
Time Frame: Insertion to Removal / maximum 3 months
Measure: Number; unit: percentage of enrolled subjects
Arm/Group | Single Arm Study
Number analyzed (Participants) | 101
percentage of enrolled subjects | 37

ADVERSE EVENTS:
Time Frame: This observationaol study included recording of line occlusions and incidence of venous thrombosis from the time of PICC insertion until removal of the PICC line or for a maximum of 90 days.
Arm/Group | Single Arm Study
Serious Adverse Events (participants affected / at risk) | 0/101
Other Adverse Events (participants affected / at risk) | 6/101
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Study (N=101)
Venous thrombosis (Blood and lymphatic system disorders) | 6 — Symptomatic venous thrombus in upper extremity ( PICC arm); verified via standard ultrasonography procedure.

LIMITATIONS AND CAVEATS:
Further comparative studies standarizing the management of PICC line flushing solutions and type if PICC line required to provide comparative and evidence based clinical practice recommendations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No